CLINICAL TRIAL: NCT05629715
Title: A Prospective, Randomized, Unblinded Trial Comparing Conventional Instrumentation, Hand-Held Accelerometer Based Computer Navigation, and Robotic Assistance Techniques in Total Knee Arthroplasty
Brief Title: Conventional Instrumentation, Computer Navigation, and Robotic Assistance Techniques in TKA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decision
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Erik N. Zeegen, MD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#21-002140
Record Dates: First submitted 2022-08-24; First posted 2022-11-29 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A maximum of 300 subjects in each arm (900 total) are to be enrolled in this study. In order to minimize selection bias, the surgeon will randomize the instrumentation technique used. Randomization will be accomplished via a random number generator in Microsoft Excel in a 1:1:1 ratio. The patient will know which treatment arm they are in at the time of study consent. They will be ineligible for the study if they ask to change treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- ROSA (Active Comparator): Subjects randomly assigned to this arm will undergo a primary total knee arthroplasty procedure using the ROSA Knee System.
  Interventions: Device: ROSA Knee System
- KneeAlign (Active Comparator): Subjects randomly assigned to this arm will undergo a primary total knee arthroplasty procedure using the KneeAlign navigation system.
  Interventions: Device: KneeAlign Computer Assisted Navigation System
- Conventional (No Intervention): Subjects randomly assigned to this arm will undergo a primary total knee arthroplasty procedure using conventional instrumentation.

INTERVENTIONS:
Device: ROSA Knee System — The Zimmer Biomet ROSA Knee System is a commercially available, FDA approved robotic assistant for performing TKA. It uses preoperative x-rays to create a three-dimensional image of the patient's knee anatomy which is used to create a preoperative template of the implants to be used and provides intraoperative guidance for bone cuts during the TKA. The robotic system also assesses the soft tissue envelope around the knee and can assist with the soft tissue balancing of the knee arthroplasty. Alternatively, it can also be used in an imageless mode where bone cuts are performed based on intra-operative mapping using anatomic landmarks.
  Arms: ROSA
Device: KneeAlign Computer Assisted Navigation System — The OrthAlign KneeAlign computer assisted navigation system is a commercially available device that uses gyroscopic limb position sensing technology mounted to intramedullary and extramedullary jigs to measure bone resection cuts in TKA that ultimately dictate implant position.
  Arms: KneeAlign

SUMMARY:
Knee osteoarthritis is a debilitating disease that can cause severe knee pain and significant limitations to patients' activities of daily living. Total knee arthroplasty (TKA), also known as knee replacement surgery, is a well-established and successful procedure for treatment of end-stage knee osteoarthritis. Over the years, TKA surgical techniques and implant technology have improved, resulting in better patient outcomes and implant survivorship. Despite continuous improvements being made to this high demand procedure, malalignment of component position is a well-known cause of post-operative complications, including knee pain, component loosening, and failure requiring revision surgery.

Advanced techniques that utilize computer navigation or robotic-arm assistance have been developed in an attempt to avoid malalignment. Both technologies were created with the goal of improving the precision of implant positioning and implant sizing in order to improve lower limb alignment and joint line alignment. The OrthoAlign KneeAlign computer assisted navigation system is a commercially available device that uses gyroscopic limb position sensing technology mounted to intramedullary and extramedullary jigs to measure bone resection cuts in TKA that ultimately dictate implant position. The Zimmer Biomet ROSA Knee System is a commercially available, FDA-approved robotic assistant for performing TKA. It uses pre-operative x-rays to create a three-dimensional image of the patient's knee anatomy, which is used to create a pre-operative template of the implants to be used and provides intra-operative guidance for bone cuts during the TKA. The robotic system also assesses the soft tissue envelope around the knee and can assist with the soft tissue balancing of the knee arthroplasty. Alternatively, it can also be used in an imageless mode where bone cuts are performed based on intra-operative mapping using anatomic landmarks. To date, there have been no prospective studies comparing the implant positioning and patient outcomes directly of the KneeAlign system with the ROSA system and conventional TKA instrumentation techniques.

DETAILED DESCRIPTION:
This is a prospective, single center, unblinded, randomized clinical study designed to facilitate the collection and evaluation of workflow efficiency, patient pain and function, adverse event data, and radiographic outcomes for patients undergoing TKA with one of three instrumentation techniques. This clinical study will include Persona and Legion product families using the ROSA Knee System, KneeAlign navigation system, or conventional instrumentation.

The primary objective of this study is to collect and compare clinical and surgical data using the commercially available ROSA Knee System instrumentation or OrthAlign KneeAlign system compared with conventional TKA instrumentation. The hypothesis is that the ROSA Knee System and KneeAlign system will demonstrate greater accuracy and more consistent component position and greater patient reported outcome scores compared to conventional TKA surgery. The investigators suspect that the ROSA system may be more accurate and precise than the KneeAlign system.

A maximum of 300 subjects in each arm (900 total) are to be enrolled in this study. In order to minimize selection bias, the investigator will randomize the instrumentation technique used. Randomization will be accomplished via a random number generator in a 1:1:1 ratio. The subject will know which treatment arm they are in at the time of study consent. They will be ineligible for the study if they ask to change treatment arms. The Principal Investigator and Co-Investigators will be skilled in TKA and experienced implanting Persona or Legion TKA system. Two of the investigators will only be using the Persona TKA system as this is their current standard of practice. One of the other investigators will use the Legion TKA system as this is their standard of practice. In order to avoid potential selection bias, each investigator will offer study participation to each consecutive eligible patient presenting as a candidate for primary TKA using the aforementioned implants. All study subjects will undergo preoperative clinical evaluations prior to their TKA.

An a priori power analysis was conducted using G*Power 3.1 Data Analysis program to determine the sample size based on a Cohen's f-statistic of 0.25. Power was set at 0.95 and with an alpha of 0.05. Total sample size based on these parameters was 252 patients. Considering that three surgeons, who perform approximately 250 TKAs per year each, will be involved, the investigators estimate that an ability to enroll approximately one-third of all eligible patients seeking TKA and, thus, set a goal for 300 patients to account for patient attrition after study initiation.

Through the use of either conventional, computer navigated or robotic techniques, standard operating procedures will be followed and all surgical procedures will be performed under aseptic conditions. Investigators will implant all commercially available components in compliance with corresponding labeling requirements, and in accordance with appropriate surgical technique(s).

Post-surgical management for study subjects will follow the investigator's standard of care for patients undergoing TKA (e.g., prophylactic antibiotic therapy, prevention of deep vein thrombosis, prevention of pulmonary embolism, etc.). Post-surgical rehabilitative therapy will be as prescribed by the investigator. Post-operative clinical evaluation will be conducted at approximately 6 weeks, 3 months, 6 months and 1 year post-operatively. Subjects will be followed post-operatively for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a minimum of 18 years of age
* Independent of study participation, patient is a candidate for commercially available Persona or Legion knee components implanted in accordance with product labeling
* Patient has participated in this study-related Informed Consent process
* Patient is willing and able to provide written Informed Consent by signing and dating the Institutional Review Board (IRB) or Ethics Committee (EC) approved Informed Consent form
* Patient is willing and able to complete scheduled study procedures and follow-up evaluations

Exclusion Criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies
* Patient has undergone contralateral unicompartmental knee arthroplasty (UKA) or total knee arthroplasty (TKA) within the last 18 months
* Hip pathology with significant bone loss (e.g., avascular necrosis of the femoral head with collapse, severe dysplasia of the femoral head or the acetabulum)
* Hip pathology severely limiting range of motion (e.g., arthrodesis, severe contracture, chronic severe dislocation)
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.)
* Patient has previously received partial or total knee arthroplasty for the ipsilateral knee
* Patients with active knee joint infections (determined clinically at time of pre-op evaluation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Implant Positioning | Pre-Op
  Radiographic evaluation of post-operative implant positioning compared to pre-operative planning.
Implant Positioning | Up to 6 Hours
  Radiographic evaluation of post-operative implant positioning compared to pre-operative planning.
Implant Positioning | 6 weeks
  Radiographic evaluation of post-operative implant positioning compared to pre-operative planning.
Implant Positioning | 3 months
  Radiographic evaluation of post-operative implant positioning compared to pre-operative planning.
Implant Positioning | 6 months
  Radiographic evaluation of post-operative implant positioning compared to pre-operative planning.
Implant Positioning | 1 year
  Radiographic evaluation of post-operative implant positioning compared to pre-operative planning.

SECONDARY OUTCOMES:
Knee Questionnaire | Pre-Op
  Forgotten Joint Score - 12 questions scored 1 (never) to 5 (mostly). The 12 scores are aggregated to a raw score from 12-60. This raw score is linearly transformed to a 0-100 scale and then reversed to obtain a final score. A high final score indicates a good outcome.
Knee Outcome Score | Pre-Op
  Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) - 7 questions scored from 0 (none) to 4 (extreme). The 7 scores are aggregated to a score from 0-28 which inversely equates to an interval score of 0-100. An interval score of 0 equates to total knee disability and an interval score of 100 indicates perfect knee health.
Health Questionnaire | Pre-Op
  EuroQol-5 Dimensions-5 Level (EQ-5D-5L) - This consists of a descriptive system and a visual analogue scale (VAS). The descriptive system comprises five questions, scored 1 (no problems) to 5 (extreme problems). The score for each question can be combined into a 5-digit number that describes the patient's health state. A score of 11111 would be optimal. A score of 55555 would equate to complete disability. The VAS is a self-rated vertical scale, from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine").
Objective Knee Assessment | Pre-Op
  Charnley Functional Classification - An objective knee indicator with 6 possible classifications: Unilateral Knee Arthritis; Unilateral Total Knee Arthroplasty (TKA), opposite knee arthritic; Bilateral TKA; TKA, but remote arthritis affecting ambulation; TKA, but medical condition affecting ambulation; Unilateral or Bilateral TKA with unilateral or bilateral Total Hip Arthroplasty.
Knee Alignment | Pre-Op
  Anatomic alignment measured on Anterior Posterior (AP) Standing x-ray
Knee Instability Medial/Lateral (M/L) | Pre-Op
  M/L instability measured in full extension
Knee Instability Anterior/Posterior (A/P) | Pre-Op
  A/P instability measured at 90 degrees
Joint Motion | Pre-Op
  Knee Range of Motion measured in degrees
Knee Questionnaire | 6 weeks
  Forgotten Joint Score - 12 questions scored 1 (never) to 5 (mostly). The 12 scores are aggregated to a raw score from 12-60. This raw score is linearly transformed to a 0-100 scale and then reversed to obtain a final score. A high final score indicates a good outcome.
Knee Outcome Score | 6 weeks
  KOOS, JR. - 7 questions scored from 0 (none) to 4 (extreme). The 7 scores are aggregated to a score from 0-28 which inversely equates to an interval score of 0-100. An interval score of 0 equates to total knee disability and an interval score of 100 indicates perfect knee health.
Health Questionnaire | 6 weeks
  EQ-5D-5L - This consists of a descriptive system and a visual analogue scale (VAS). The descriptive system comprises five questions, scored 1 (no problems) to 5 (extreme problems). The score for each question can be combined into a 5-digit number that describes the patient's health state. A score of 11111 would be optimal. A score of 55555 would equate to complete disability. The VAS is a self-rated vertical scale, from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine").
Objective Knee Assessment | 6 weeks
  Charnley Functional Classification - An objective knee indicator with 6 possible classifications: Unilateral Knee Arthritis; Unilateral Total Knee Arthroplasty (TKA), opposite knee arthritic; Bilateral TKA; TKA, but remote arthritis affecting ambulation; TKA, but medical condition affecting ambulation; Unilateral or Bilateral TKA with unilateral or bilateral Total Hip Arthroplasty.
Knee Alignment | 6 weeks
  Anatomic alignment measured on AP Standing x-ray
Knee Instability M/L | 6 weeks
  M/L instability measured in full extension
Knee Instability A/P | 6 weeks
  A/P instability measured at 90 degrees
Joint Motion | 6 weeks
  Knee Range of Motion measured in degrees
Patellar Tracking | 6 weeks
  Investigator assessment of any abnormalities in patellar tracking post-operatively
Patient Satisfaction | 6 weeks
  Question to be completed by the subject indicating their level of satisfaction with the operated knee as either Very Satisfied, Satisfied, Uncertain, or Unsatisfied.
Knee Questionnaire | 3 months
  Forgotten Joint Score - 12 questions scored 1 (never) to 5 (mostly). The 12 scores are aggregated to a raw score from 12-60. This raw score is linearly transformed to a 0-100 scale and then reversed to obtain a final score. A high final score indicates a good outcome.
Knee Outcome Score | 3 months
  KOOS, JR. - 7 questions scored from 0 (none) to 4 (extreme). The 7 scores are aggregated to a score from 0-28 which inversely equates to an interval score of 0-100. An interval score of 0 equates to total knee disability and an interval score of 100 indicates perfect knee health.
Health Questionnaire | 3 months
  EQ-5D-5L - This consists of a descriptive system and a visual analogue scale (VAS). The descriptive system comprises five questions, scored 1 (no problems) to 5 (extreme problems). The score for each question can be combined into a 5-digit number that describes the patient's health state. A score of 11111 would be optimal. A score of 55555 would equate to complete disability. The VAS is a self-rated vertical scale, from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine").
Objective Knee Assessment | 3 months
  Charnley Functional Classification - An objective knee indicator with 6 possible classifications: Unilateral Knee Arthritis; Unilateral Total Knee Arthroplasty (TKA), opposite knee arthritic; Bilateral TKA; TKA, but remote arthritis affecting ambulation; TKA, but medical condition affecting ambulation; Unilateral or Bilateral TKA with unilateral or bilateral Total Hip Arthroplasty.
Knee Alignment | 3 months
  Anatomic alignment measured on AP Standing x-ray
Knee Instability M/L | 3 months
  M/L instability measured in full extension
Knee Instability A/P | 3 months
  A/P instability measured at 90 degrees
Joint Motion | 3 months
  Knee Range of Motion measured in degrees
Patellar Tracking | 3 months
  Investigator assessment of any abnormalities in patellar tracking post-operatively
Patient Satisfaction | 3 months
  Question to be completed by the subject indicating their level of satisfaction with the operated knee as either Very Satisfied, Satisfied, Uncertain, or Unsatisfied.
Knee Questionnaire | 6 months
  Forgotten Joint Score - 12 questions scored 1 (never) to 5 (mostly). The 12 scores are aggregated to a raw score from 12-60. This raw score is linearly transformed to a 0-100 scale and then reversed to obtain a final score. A high final score indicates a good outcome.
Knee Outcome Score | 6 months
  KOOS, JR. - 7 questions scored from 0 (none) to 4 (extreme). The 7 scores are aggregated to a score from 0-28 which inversely equates to an interval score of 0-100. An interval score of 0 equates to total knee disability and an interval score of 100 indicates perfect knee health.
Health Questionnaire | 6 months
  EQ-5D-5L - This consists of a descriptive system and a visual analogue scale (VAS). The descriptive system comprises five questions, scored 1 (no problems) to 5 (extreme problems). The score for each question can be combined into a 5-digit number that describes the patient's health state. A score of 11111 would be optimal. A score of 55555 would equate to complete disability. The VAS is a self-rated vertical scale, from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine").
Knee Questionnaire | 1 year
  Forgotten Joint Score - 12 questions scored 1 (never) to 5 (mostly). The 12 scores are aggregated to a raw score from 12-60. This raw score is linearly transformed to a 0-100 scale and then reversed to obtain a final score. A high final score indicates a good outcome.
Knee Outcome Score | 1 year
  KOOS, JR. - 7 questions scored from 0 (none) to 4 (extreme). The 7 scores are aggregated to a score from 0-28 which inversely equates to an interval score of 0-100. An interval score of 0 equates to total knee disability and an interval score of 100 indicates perfect knee health.
Health Questionnaire | 1 year
  EQ-5D-5L - This consists of a descriptive system and a visual analogue scale (VAS). The descriptive system comprises five questions, scored 1 (no problems) to 5 (extreme problems). The score for each question can be combined into a 5-digit number that describes the patient's health state. A score of 11111 would be optimal. A score of 55555 would equate to complete disability. The VAS is a self-rated vertical scale, from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine").
Objective Knee Assessment | 1 year
  Charnley Functional Classification - An objective knee indicator with 6 possible classifications: Unilateral Knee Arthritis; Unilateral Total Knee Arthroplasty (TKA), opposite knee arthritic; Bilateral TKA; TKA, but remote arthritis affecting ambulation; TKA, but medical condition affecting ambulation; Unilateral or Bilateral TKA with unilateral or bilateral Total Hip Arthroplasty.
Knee Alignment | 1 year
  Anatomic alignment measured on AP Standing x-ray
Knee Instability M/L | 1 year
  M/L instability measured in full extension
Knee Instability A/P | 1 year
  A/P instability measured at 90 degrees
Joint Motion | 1 year
  Knee Range of Motion measured in degrees
Patellar Tracking | 1 year
  Investigator assessment of any abnormalities in patellar tracking post-operatively
Patient Satisfaction | 1 year
  Question to be completed by the subject indicating their level of satisfaction with the operated knee as either Very Satisfied, Satisfied, Uncertain, or Unsatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Santa Monica Medical Center, Santa Monica, California, United States